CLINICAL TRIAL: NCT01398683
Title: Comparison Epidural Anesthesia and General Anesthesia in Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201104080RC
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2011-07

CONDITIONS: Epidural Anesthesia; Laparoscopic Cholecystectomy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Comparison of epidural anesthesia and general anesthesia for laparoscopic cholecystectomy, patients in the surgery and the effectiveness of anesthesia after surgery, the incidence of side effects or complications, and postoperative recovery of the body of the differences

ELIGIBILITY:
Inclusion Criteria:

* Underwent laparoscopic cholecystectomy in patients

Exclusion Criteria:

* Unconsciousness or can not express their own feelings of the patient

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Underwent laparoscopic cholecystectomy in patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Estimated); Study Completion 2014-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yao Ming Wu, Bachelor, Principal Investigator — National Taiwan University Hospital